CLINICAL TRIAL: NCT01403688
Title: Effects of Controlled Ovarian Hyperstimulation (COH) With Letrozole and Gonadotropin in Women at High Risk for Breast Cancer
Brief Title: Effects of Controlled Ovarian Hyperstimulation (COH) With Letrozole and Gonadotropin
Status: Completed | Type: Observational
Sponsor: University of Kansas (Other)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 11357
Record Dates: First submitted 2011-07-14; First posted 2011-07-27 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Infertility; Breast Cancer
Keywords: fertility high risk, controlled ovarian stimulation, breast cancer
MeSH Terms: conditions — Infertility; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Random Fine Needle Aspiration (RPFNA): RPFNA
  Interventions: Procedure: RPFNA

INTERVENTIONS:
Procedure: RPFNA — 1. Baseline RPFNA within 3 month prior to the initial COH cycle or within the first 10 days of the treatment cycle (delete this).
  2. Repeat RPFNA if pregnancy is not achieved: 6 to 18 months following baseline assessment
  3. Repeat RPFNA if pregnancy is achieved: approximately 12 months after discontinuation of breast feeding

SUMMARY:
Fertility drugs have the effect of increasing hormone levels. Higher hormone levels from infertility treatments may increase breast cancer risk, but there has not been enough research to know for sure. Researchers want to use a method of taking breast tissue cells from women who are having infertility treatment. The breast tissue cells might show changes that would indicate an increased risk of cancer. The method of taking the breast tissue cells is called Fine Needle Aspiration (FNA).

The purpose of this study is to examine the changes in breast tissue, in women at high risk of breast cancer who are being treated with controlled ovarian hyperstimulation.

ELIGIBILITY:
Inclusion criteria:

1. Women must be at increased risk for breast cancer based on any of the following criteria:

   * Age 30 or older with no prior live birth.
   * Mutations associated with hereditary cancer (BRCA1 or 2, P53, PTEN)
   * Family history of breast cancer including one first degree or multiple second degree relatives
   * History of chest radiation before age 30
   * Multiple prior breast biopsies
   * Precancerous conditions (DCIS, LCIS, AH)
   * Prior history of breast or ovarian cancer
   * Estimated mammographic breast density > 50%
2. Must be undergoing infertility treatment at the University of Kansas with Controlled Ovarian Hyper-stimulation (COH)
3. Must be between the ages of 21-45 (both inclusive) with Day 3 FSH less than 12 IU/L, Day 3 E2 less than 80 pg/ml

Exclusion criteria:

1. Women under 21 or over 45 years old
2. Day 3 FSH over 12 IU/L, Day 3 E2 over 80 pg/ml
3. Women who do not meet risk criteria above
4. History of hypersensitivity to letrozole or gonadotropin
5. Uterine and adnexal pathology
6. Use of clomid or gonadotropin within 30days before the letrozole cycle
7. Any severe chronic disease of relevance for reproductive function

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infertility Patients undergoing COH treatment and at high risk for breast cancer
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2011-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
evaluation with pre- and post-treatment(COH) breast cytomorphometry and biomarkers | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Kim, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States